CLINICAL TRIAL: NCT03813953
Title: The Effect of Analgesic Modalities on Long Term Outcomes Following Open Liver Resection
Acronym: LIVER 3
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Edinburgh (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 258352
Record Dates: First submitted 2018-12-10; First posted 2019-01-23 (Actual); Last update posted 2024-05-22 (Actual); Status verified 2024-05

CONDITIONS: Liver Cancer
MeSH Terms: conditions — Liver Neoplasms | interventions — Hepatectomy

STUDY DESIGN:
Intervention Model Description: Long term follow up of previously randomised populations.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Local Anaesthetic Wound Infiltration (Experimental): Wound catheter delivering local anaesthetic for 48 hours post-operatively following liver resection
  Interventions: Procedure: Liver resection
- Epidural (Active Comparator): Conventional practice following liver resection
  Interventions: Procedure: Liver resection

INTERVENTIONS:
Procedure: Liver resection — Resection of diseased liver

SUMMARY:
The LIVER (Local Infiltration Versus Epidural after Liver Resection) and LIVER 2 (Local Infiltration Versus Epidural after Liver Resection 2) studies were randomised controlled trials that compared epidural analgesia with local anaesthetic wound infiltration as post-operative analgesia in patients undergoing open liver resection.

The overall findings of this trial were of similar rates of morbidity and pain control post-operatively but a reduced recovery time for the wound catheter group. As a result, wound catheter local anesthetic infiltration has become increasingly utilized in this unit and within other units throughout the country and worldwide.

Epidural use has been associated with improved long term outcomes following abdominal cancer surgery. This study is therefore a long term follow up study of the LIVER and LIVER 2 trials to assess survival between the two groups.

DETAILED DESCRIPTION:
The LIVER and LIVER 2 studies were randomised controlled trials that compared epidural analgesia with local anaesthetic wound infiltration as post-operative analgesia in patients undergoing open liver resection.

The overall findings of this trial were of similar rates of morbidity and pain control post-operatively but a reduced recovery time for the wound catheter group. As a result, wound catheter local anesthetic infiltration has become increasingly utilized in this unit and within other units throughout the country and worldwide.

There has been some evidence however, that epidural analgesia post-operatively can have a positive impact on long term survival in patients undergoing abdominal surgery for cancer. The reasons for this are not well established but it is proposed that the protective effect against the immunosuppression following major surgery that epidural has can aid in the cancer prevention process. There remains no randomised controlled trials looking at this subject in open liver surgery.

The aim of this study is to assess the overall and disease free survival of the patients who participated in the LIVER and LIVER 2 trials.

The primary outcome is 5 year overall survival. Data will be observed from electronic (or non electronic) patient records, information and statistics department data and general practice records as required.

Overall survival at 1 and 3 years Disease free survival at 1, 3 and 5 years (Data will be observed from Lothian hepatobiliary multi-disciplinary team meeting data and follow up CT/MRI scan dates)

Median overall and disease free survival Survival according to individual pathology subgroups.

Participants will be identified from study records of the LIVER and LIVER 2 trials. This will be performed by the two study investigators.

ELIGIBILITY:
Inclusion Criteria:

* Patients who participated in the LIVER and LIVER 2 trials who had diagnoses of a malignancy and underwent liver resection for this malignancy.

Exclusion Criteria:

* Patients who had liver resection for benign disease. Patients who participated in the LIVER/LIVER2 trials but who did not undergo resection.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 160 (Actual)
Dates: Start 2019-03-06 (Actual); Primary Completion 2019-08-30 (Actual); Study Completion 2019-08-30 (Actual)

PRIMARY OUTCOMES:
Overall survival in months | 5 years
  Number of months from the date of surgery to the date of death or the censor date

SECONDARY OUTCOMES:
overall survival | 3 years
  Number of months from the date of surgery to the date of death or the censor date
Disease free survival | 5 years
  Number of months from the date of surgery to the date of disease recurrence or the censor date

CONTACTS AND LOCATIONS:
Overall Officials: Michael Hughes, Principal Investigator — NHS Lothian
Locations (1):
- NHS Lothian, Edinburgh, United Kingdom

IPD SHARING:
Plan to Share IPD: No